CLINICAL TRIAL: NCT05176782
Title: Randomized Clinical Trial: Comparison Between Histidine-tryptophan-ketoglutarate Cardioplegia and Cold Blood Cardioplegia for Myocardial Protection for Fallot Tetralogy Patients Undergoing Total Repair
Brief Title: Comparison Between Histidine-tryptophan-ketoglutarate Cardioplegia and Cold Blood Cardioplegia for Myocardial Protection for Fallot Tetralogy Patients Undergoing Total Repair
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, samar mohammed, Lecturer of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FAMSU R 206/2021
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (HTK cardioplegia) (Active Comparator): will receive HTK cardioplegia in volume 30 ml/Kg given by antegrade route through an aortic route cannula.
  Interventions: Drug: HTK cardioplegia
- Group B ( Cold Cardioplegia) (Active Comparator): will receive group cold Blood Cardioplegia in volume 20mL/kg given by antegrade route through an aortic route cannula and repeated 10mL/kg/dose every 25minutes at 8-12°C for maintenance. This technique considered the standard management in this age.
  Interventions: Drug: Cold Cadioplegia

INTERVENTIONS:
Drug: HTK cardioplegia — will receive HTK cardioplegia in volume 30 ml/Kg given by antegrade route through an aortic route cannula.
  Arms: Group A (HTK cardioplegia)
Drug: Cold Cadioplegia — as the will receive group cold Blood Cardioplegia in volume 20mL/kg given by antegrade route through an aortic route cannula and repeated 10mL/kg/dose every 25minutes at 8-12°C for maintenance. This technique considered the standard management in this age.
  Arms: Group B ( Cold Cardioplegia)

SUMMARY:
Randomized clinical trial: comparison between Histidine-tryptophan-ketoglutarate cardioplegia and cold blood cardioplegia for myocardial protection for Fallot tetralogy patients undergoing total repair This study aims to compare HTK cardioplegic solution and cold blood cardioplegia to provide optimal myocardial protection for a patient with tetralogy of Fallot planned for total repair.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with tetralogy of Fallot spectrum.
* Sex (males and females)
* Age 6 months- 5 years.

Exclusion Criteria:

* Persistent left SVC draining in the coronary sinus.
* Mental or neurologic disorders.
* Preoperative critically ill patients.
* Parents or legal guardian refusal.
* Fallot repair with transannular patch( as it will affect on the RV function as a single agent after reperfusion)

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
• Vasoactive-Inotropic Score | From time of separation of cardioplumonary bypass till 24 hours post operative
  Calculate the doses of vasoactive drugs used

CONTACTS AND LOCATIONS:
Locations (1):
- Samar Soliman, Cairo, Nasr City, Egypt